CLINICAL TRIAL: NCT05933486
Title: A Multicenter, Randomized, Double-blind Study on the Efficacy and Safety of Tongluo-Kaibi Tablet in the Treatment of Fibromyalgia Syndrome
Brief Title: Efficacy and Safety of Tongluo-Kaibi Tablet in Patients With Fibromyalgia Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Quan Jiang (Other)
Responsible Party: Sponsor-Investigator, Quan Jiang, chief physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Organization: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022013P7A02
Record Dates: First submitted 2023-06-28; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Fibromyalgia Syndrome
Keywords: Tongluo-Kaibi Tablet; Traditional Chinese Medicine; Fibromyalgia Syndrome
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tongluo-Kaibi tablet plus placebo of pregabalin (Experimental)
  Interventions: Drug: Tongluo-Kaibi tablet plus placebo of pregabalin
- placebo of Tongluo-Kaibi tablet plus pregabalin (Active Comparator)
  Interventions: Drug: placebo of Tongluo-Kaibi tablet plus pregabalin

INTERVENTIONS:
Drug: Tongluo-Kaibi tablet plus placebo of pregabalin — Tongluo-Kaibi Tablet 0.93g qd； Placebo of pregabalin 150mg qd. If the patient can tolerate it, it will be increased to 150mg bid one week later. If the patient cannot tolerate it, it will be maintained at 150mg qd until the 8th week.
  Arms: Tongluo-Kaibi tablet plus placebo of pregabalin
Drug: placebo of Tongluo-Kaibi tablet plus pregabalin — placebo of Tongluo-Kaibi Tablet 0.93g qd； Pregabalin 150mg qd. If the patient can tolerate it, it will be increased to 150mg bid one week later. If the patient cannot tolerate it, it will be maintained at 150mg qd until the 8th week.
  Arms: placebo of Tongluo-Kaibi tablet plus pregabalin

SUMMARY:
This study is a multi-center, randomized, double-blinded, controlled trial with two parallel arms. The aim of the study is to evaluate efficacy and safety of Tongluo-Kaibi tablets in patients with Fibromyalgia Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Those who meet the classification criteria for Fibromyalgia formulated by the American Rheumatology Association in 2016.
* Pain VAS score ≥ 4 points.
* The variety and dosage of the medication used to treat the disease should be stable for at least 2 weeks.

Exclusion Criteria:

* Severe cardiovascular and cerebrovascular diseases.
* Malignant tumors, hematological diseases, inflammatory arthritis, or other serious or progressive systemic diseases.
* ALT and AST are more than 2 times the upper limit of normal.
* Cr is more than 1.2 times the upper limit of normal.
* Allergic constitution or allergic to experimental drugs Tongluo-Kaibi tablet, pregabalin capsules, excipients or similar ingredients.
* Pregnant, lactating or recently planned pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-11 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
VAS | 8 weeks
  Visual Analogue Score

SECONDARY OUTCOMES:
MFI-20 | 8 weeks
  Multidimensional Fatigue Inventory
BDI | 8 weeks
  Beck Depression Inventory
PSQI | 8 weeks
  Pittsburgh Sleep Quality Index
WPI | 8 weeks
  Widespread Pain Index

IPD SHARING:
Plan to Share IPD: No